CLINICAL TRIAL: NCT02623348
Title: Use of Pedometers to Measure and Increase Walking Among Patients With ESRD
Acronym: PED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-02719
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: End-stage Renal Disease
Keywords: dialysis; end-stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pedometer (Experimental): Patients will be given pedometers and instructions to increase physical activity based on pedometer output
  Interventions: Behavioral: pedometer
- usual care (No Intervention): No intervention

INTERVENTIONS:
Behavioral: pedometer — pedometer-based physical activity recommendations
  Arms: pedometer

SUMMARY:
Randomized controlled trial using pedometers to increase physical activity among patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* on hemodialysis for ≥ 3 months
* able to walk
* able to give informed consent and willing to participate

Exclusion Criteria:

* unable to walk
* unable to understand directions or give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Sheshadri A, Kittiskulnam P, Delgado C, Sudore RL, Lai JC, Johansen KL. Association of Cognitive Function Screening Results with Adherence and Performance in a Pedometer-Based Intervention. Am J Nephrol. 2021;52(5):420-428. doi: 10.1159/000516130. Epub 2021 May 12. PMID 33979802
- [Derived] Sheshadri A, Kittiskulnam P, Delgado C, Sudore R, Lai JC, Johansen KL. Association of motivations and barriers with participation and performance in a pedometer-based intervention. Nephrol Dial Transplant. 2020 Aug 1;35(8):1405-1411. doi: 10.1093/ndt/gfaa047. PMID 32437568
- [Derived] Sheshadri A, Kittiskulnam P, Lai JC, Johansen KL. Effect of a pedometer-based walking intervention on body composition in patients with ESRD: a randomized controlled trial. BMC Nephrol. 2020 Mar 16;21(1):100. doi: 10.1186/s12882-020-01753-5. PMID 32178648
- [Derived] Sheshadri A, Kittiskulnam P, Lazar AA, Johansen KL. A Walking Intervention to Increase Weekly Steps in Dialysis Patients: A Pilot Randomized Controlled Trial. Am J Kidney Dis. 2020 Apr;75(4):488-496. doi: 10.1053/j.ajkd.2019.07.026. Epub 2019 Nov 1. PMID 31679747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from 3 local San Francisco dialysis clinics
Pre-assignment Details: Baseline assessment performed prior to random assignment
Groups:
- Pedometer: Patients will be given pedometers and weekly instructions to increase physical activity based on pedometer output over the prior week.
- Usual Care: Recommendations for physical activity as determined by American Heart Association and American College of Sports Medicine at time of enrollment only. Otherwise, usual care.
Period: Overall Study
Arm/Group | Pedometer | Usual Care
Started | 30 | 30
3-month Assessment | 27 | 26
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pedometer | Usual Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [53 to 66] | 56 [51 to 65] | 58 [53 to 65.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 28 | 19 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 14 | 11 | 25
  White | 4 | 5 | 9
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.9 [25.3 to 32.9] | 31.6 [26.7 to 34.6] | 29 [25.5 to 34.4]
Dialysis Vintage (Years) [Mean (Inter-Quartile Range); unit: years] | 3.7 [1.5 to 7.2] | 1.9 [0.95 to 4.7] | 3.1 [1.1 to 5.8]
Hemoglobin [Median (Inter-Quartile Range); unit: mg/dL] | 10.6 [9.6 to 11.7] | 10.9 [9.8 to 11.7] | 10.7 [9.8 to 11.7]
Serum Albumin [Median (Inter-Quartile Range); unit: g/dL] | 3.9 [3.7 to 4.1] | 3.9 [3.6 to 4.1] | 3.9 [3.7 to 4.1]
Standardized Kt/V [Median (Inter-Quartile Range); unit: unitless, per week] | 2.30 [2.07 to 2.44] | 2.37 [2.1 to 2.5] | 2.32 [2.09 to 2.47]
Currently smoking [Count of Participants; unit: Participants] | 6 | 3 | 9
Hypertension [Count of Participants; unit: Participants] | 28 | 28 | 56
Diabetes [Count of Participants; unit: Participants] | 10 | 12 | 22
Coronary Artery Disease [Count of Participants; unit: Participants] | 11 | 8 | 19
Congestive Heart Failure [Count of Participants; unit: Participants] | 9 | 8 | 17
Stroke [Count of Participants; unit: Participants] | 2 | 4 | 6
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 4 | 1 | 5
HIV [Count of Participants; unit: Participants] | 0 | 1 | 1
Arrhythmia [Count of Participants; unit: Participants] | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: change in steps per day from pedometer
Time Frame: Baseline and 12 weeks
Measure: Median (95% Confidence Interval); unit: steps/day
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
steps/day | 1474 [40 to 3538] | 180 [-650 to 1040]
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; p < 0.01, linear mixed modeling — Threshold for significance: <0.05

2. Secondary Outcome: Physical Performance
Description: change in score on the Short Physical Performance Battery (0-12), higher scores indicate greater physical performance
Time Frame: Baseline and 12 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
score on a scale | 0 [0 to 1] | 0 [-1 to 1]

3. Secondary Outcome: Self-reported Physical Functioning
Description: Change in score on the Physical Function scale of the Short-Form 36 Health Survey (scale from 0-100, higher numbers indicate better physical functioning)
Time Frame: Baseline and 12 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
score on a scale | 0 [-10 to 5] | 5 [-5 to 10]

4. Secondary Outcome: Change in Activities of Daily Living Score
Description: Barthel's Index of Daily Activities (Index range 0-20, higher scores indicate greater functional independence)
Time Frame: Baseline and 12 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
score on a scale | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Change in Symptom Burden on the Dialysis Symptoms Index
Description: Dialysis symptom index (symptom burden ranges from 0 - 29 symptoms experienced)
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
score on a scale | 1 [-1.5 to 2] | 0 [-2 to 2]

6. Secondary Outcome: Change in Total Body Muscle Mass (Adjusted by Height Squared)
Description: (TBMM calculated from measurements of intracellular water from bioimpedance spectrometry)
Time Frame: Baseline and 12 weeks
Population: Note: we were unable to obtain body composition measures from all participants at baseline and 12 weeks (Missing data from: 3 with metal implants, 1 with pacemaker, 2 with poor quality of measurement likely related to fluid shifts)
Measure: Median (Inter-Quartile Range); unit: kg/m2
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 23 | 24
kg/m2 | 0.30 [-0.50 to 0.76] | -0.47 [-0.90 to 0.35]

7. Secondary Outcome: Change in Endothelial Function
Description: Reactive hyperemia index (RHI) using peripheral arterial tonometry. RHI is a non-invasive measure of endothelial function, measured using the EndoPAT 2000 (Itamar Medical). The pulse amplitude in the middle fingers of both hands was recorded for five minutes. A blood pressure cuff was then inflated in one arm (which did not have a vascular access in place) to at least 60 mmHg above systolic blood pressure to achieve full occlusion (minimum 200 mmHg, maximum 300 mmHg). After occlusion for 5 minutes, the cuff was deflated, and the device recorded changes in pulse amplitude for an additional 5 minutes and calculated RHI as the ratio of the post to pre occlusion amplitude of the occluded arm relative to the post to pre occlusion amplitude of the control arm, corrected for baseline vascular tone.
Time Frame: 12 weeks
Measure: Median (95% Confidence Interval); unit: unitless
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
unitless | -0.1 [-0.3 to 0.22] | 0.1 [-0.57 to 0.28]

8. Secondary Outcome: Change in the Short From 36 Vitality Scale
Description: Short Form 36 Vitality Scale (0-100, greater values indicate increased levels of energy/decreased levels of fatigue)
Time Frame: Baseline and 12 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
score on a scale | 0 [-10 to 15] | 5 [-10 to 10]

9. Secondary Outcome: Change in SDNN (ms)
Description: Standard deviation of N-N intervals as recorded on electrocardiography waveform (ms)
Time Frame: 12 weeks
Measure: Median (95% Confidence Interval); unit: ms
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
ms | 1.54 [-6.19 to 11.57] | -0.13 [-6.95 to 2.27]

10. Secondary Outcome: Change in Symptom Severity on Dialysis Symptoms Index
Description: Symptoms range from score of 0 (Not at all bothersome) to 5 (Very Bothersome) over 29 symptoms. Score ranges from 0 - 145
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pedometer | Usual Care
Number analyzed (Participants) | 27 | 26
score on a scale | 2 [-3.5 to 13] | -1 [-9 to 9]

ADVERSE EVENTS:
Time Frame: 24 months total, 6 months per patient
Arm/Group | Pedometer | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 6/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pedometer (N=30) | Usual Care (N=30)
Fatigue (General disorders) | 6 (6) | 2 (2) — Increased fatigue/weariness

LIMITATIONS AND CAVEATS:
Outcomes reported are median change within groups with 95% confidence interval. Primary analysis is difference in change between groups using linear mixed modeling. Participants were selected only from dialysis clinics in Northern California.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02623348/Prot_SAP_000.pdf